CLINICAL TRIAL: NCT02701907
Title: Low Level of Genomic Alteration to Predict Exceptional and Unexpected Response to Targeted Therapies in Patients With Solid Tumors
Brief Title: EXPRESS: EXcePtional RESponSe - Exceptional and Unexpected Response to Targeted Therapies
Acronym: EXPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UC-0105/1508; 2015-A01500-49 (Registry Identifier: ANSM)
Record Dates: First submitted 2016-01-27; First posted 2016-03-08 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Cancers
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- breast cancer (Other): In this study, we aim to assess whether tumors characterized by a low level of genomic alterations (mutation, amplification or deletion) are associated with unexpected and exceptional responses across targeted anticancer therapies. We will focus our analyses on tumor types for which molecular targeted anticancer agents are frequently prescribed
  Interventions: Other: Blood sampling
- non-small cell lung cancer (Other): In this study, the investigators aim to assess whether tumors characterized by a low level of genomic alterations (mutation, amplification or deletion) are associated with unexpected and exceptional responses across targeted anticancer therapies.
  The investigators will focus analyses on tumor types for which molecular targeted anticancer agents are frequently prescribed
  Interventions: Other: Blood sampling
- kidney cancer (Other): In this study, the investigators aim to assess whether tumors characterized by a low level of genomic alterations (mutation, amplification or deletion) are associated with unexpected and exceptional responses across targeted anticancer therapies. the investigators will focus analyses on tumor types for which molecular targeted anticancer agents are frequently prescribed
  Interventions: Other: Blood sampling
- colorectal cancer (Other): In this study, the investigators aim to assess whether tumors characterized by a low level of genomic alterations (mutation, amplification or deletion) are associated with unexpected and exceptional responses across targeted anticancer therapies. the investigators will focus analyses on tumor types for which molecular targeted anticancer agents are frequently prescribed
  Interventions: Other: Blood sampling
- ovarian cancer (Other): In this study, the investigators aim to assess whether tumors characterized by a low level of genomic alterations (mutation, amplification or deletion) are associated with unexpected and exceptional responses across targeted anticancer therapies. the investigators will focus analyses on tumor types for which molecular targeted anticancer agents are frequently prescribed
  Interventions: Other: Blood sampling
- skin cutaneous melanoma (Other): In this study, the investigators aim to assess whether tumors characterized by a low level of genomic alterations (mutation, amplification or deletion) are associated with unexpected and exceptional responses across targeted anticancer therapies. the investigators will focus analyses on tumor types for which molecular targeted anticancer agents are frequently prescribed
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling

SUMMARY:
Adult patients with metastatic or locally advanced solid malignancies (including but not limited to breast, cancer, lung adenocarcinoma or squamous cell carcinoma, colorectal cancer, ovarian cancer, renal clear cell cancer, skin cutaneous melanoma), presenting or having presented an exceptional and unexpected response to an antineoplastic targeted therapy.

DETAILED DESCRIPTION:
The primary endpoint is the rate of patients with tumors harboring a low level of genomic alteration (mutation, amplification or deletion) in genes (i.e. mutation, amplification, deletion) identified as causally implicated in cancer. A low level of genomic alteration is defined by the presence of less than the 5th quantile of genomic alterations to be expected in the given tumor type. Conversely, a high level of genomic alteration is defined by the presence of more than the 5th quantile of genomic alterations to be expected in the given tumor type.

The list of genes for which alterations are identified as causally implicated in cancer is defined by the Cancer Gene Census. This is an ongoing effort to catalogue those genes for which mutations, amplifications or deletions have been causally implicated in cancer. It is constantly updated by the Wellcome Trust Sanger Institute (UK) and available at: http://cancer.sanger.ac.uk/census (n=571 genes in September 2015)

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient ( ≥18 years old at diagnosis).
2. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.
3. Patient suffering from the following tumor type: breast cancer, lung adenocarcinoma or squamous cell carcinoma, colorectal cancer, ovarian cancer, renal clear cell cancer, skin cutaneous melanoma.
4. Metastatic or locally advanced disease.
5. Currently or previously treated with an anticancer targeted therapy in monotherapy. Targeted therapies combined with other agents are accepted only if 1/ the tumor was previously proven to be progressive under the same agents or 2/ the response or the stability has been maintained with the targeted therapy alone after the agent has been stopped.
6. Exceptional and unexpected tumor response to any marketed targeted therapy confirmed by the college of experts and defined as: complete response or partial response lasting more than six months, and not expected in more than 10% of the patients in this drug organ situation.
7. Availability and required quality of the tumor biopsy (FFPE or frozen sample) allowing for the whole exome sequencing analysis. Tumor biopsies obtained just before the initiation of the targeted therapy are preferred; otherwise any prior sample is possible.
8. Availability of normal tissue along with the tumor tissue, otherwise blood sample in order to extract constitutional DNA.

Exclusion Criteria:

1. Pediatric patient (<18 years old at diagnosis).
2. Hematological malignancy or solid tumors, which are not in the scope of tumor types described in the inclusion criteria.
3. Tumor sample not available or not reaching the required quality for whole exome sequencing analysis.
4. Absence of confirmation of the exceptional and unexpected pattern of response by the college of experts as defined above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2022-04-17 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the rate of patients with tumors harboring a low level of genomic alteration (mutation, amplification or deletion) in genes (i.e. mutation, amplification, deletion) identified as causally implicated in cancer | 42 months

SECONDARY OUTCOMES:
The secondary endpoint is the rate of tumors with low level of genomic alterations between the EXPRESS cohort and control cohorts of patients. | 42 months
Exploratory analyses will be performed to compare the profiles between the EXPRESS and the control cohorts of patients, to identify novel candidate somatic molecular profiles | 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ferté, MD PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (36):
- France (36):
  - Clinique de l'Europe, Amiens
  - CHU d'Angers, Angers
  - Institut de Cancérologie de l'Ouest (site Paul Papin), Angers
  - Centre Hospitalier Annecy Genevois (CHANGE) - site d'Annecy, Annecy
  - CHU d'Auxerre, Auxerre
  - Institut Sainte-Catherine, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hôpital Privé Sainte Marie, Chalon-sur-Saône
  - Centre Hospitalier Metropole Savoie, Chambéry
  - Centre Jean Perrin, Clermont-Ferrand
  - CH Sud Francilien, Corbeil
  - Centre Georges-François Leclerc, Dijon
  - Hôpital Privé Drôme Ardèche - Clinique Pasteur, Guilherand-Granges
  - Centre Oscar Lambret, Lille
  - CH de Longjumeau, Longjumeau
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Nord, Marseille
  - Institut Paoli-Calmettes, Marseille
  - Hôpital Clinique Claude Bernard, Metz
  - Institut de Cancérologie de Lorraine, Nancy
  - Institut de Cancérologie de l'Ouest (site René Gauducheau), Nantes
  - Centre Antoine Lacassagne, Nice
  - CHR d'Orléans - Hôpital de la Source, Orléans
  - Curie Paris, Paris
  - Hôpital Européen Georges Pompidou (HEGP), Paris
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud - Hospices Civils de Lyon, Pierre-Bénite
  - CHU de Poitiers - Pôle régional de Cancérologie, Poitiers
  - Centre Eugène Marquis, Rennes
  - Hôpitaux Drôme-Nord- Site de Romans sur Isère, Romans-sur-Isère
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No